CLINICAL TRIAL: NCT05181566
Title: Metal Ion Levels in Total Hip Arthroplasty (THA) With Modular Dual Mobility (MDM) Cup Compared to Conventional Total Hip Arthroplasty (THA) - A Multicenter Prospective Randomized Controlled Study
Brief Title: Metal Ion Levels in Total Hip Arthroplasty (THA) With Modular Dual Mobility Cup Compared to Conventional THA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Stryker Korea Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019GR0112
Record Dates: First submitted 2021-12-03; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-03

CONDITIONS: Femur Neck Fracture; Arthroplasty Complications
Keywords: Total hip arthroplasty; Metal ion; Dual mobility; Total hip replacement
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Modular dual mobility group (Experimental): A group of patients who underwent total hip replacement arthroplasty using a modular dual mobility cup
  Interventions: Procedure: Total hip replacement arthroplasty using modular dual mobility cup
- Conventional group (Active Comparator): A group of patients who underwent total hip replacement arthroplasty using a conventional acetabular cup
  Interventions: Procedure: Total hip replacement arthroplasty using conventional acetabular cup

INTERVENTIONS:
Procedure: Total hip replacement arthroplasty using modular dual mobility cup — In a total hip replacement (also called total hip arthroplasty), the damaged bone and cartilage is removed and replaced with prosthetic components
  Arms: Modular dual mobility group
Procedure: Total hip replacement arthroplasty using conventional acetabular cup — In a total hip replacement (also called total hip arthroplasty), the damaged bone and cartilage is removed and replaced with prosthetic components
  Arms: Conventional group

SUMMARY:
After total hip arthroplasty using an 'Modular Dual Mobility' acetabular cup, which is effective in reducing the risk of dislocation, one of the serious complications occurring after total hip arthroplasty, the blood metal ion concentration was compared with that of conventional total hip arthroplasty patients. This is a multicenter prospective randomized comparative study.

DETAILED DESCRIPTION:
Dislocation after total hip arthroplasty is a very serious complication not only for the patient but also for the operator, and is the second most common complication after joint dissociation. The incidence of dislocation after conventional total hip arthroplasty has been reported to be about 0.2 to 7%, and the frequency is higher in elderly patients with hip fractures and has been reported up to about 9%. In patients at high risk of dislocation, total hip arthroplasty using a dual mobility acetabular cup has the effect of reducing the risk of dislocation, and its use has been increasing in recent years. The dual mobility acetabular cup used in this study was developed in a form that can be screwed through the acetabular cup to compensate for the shortcomings of the dual mobility acetabular cup used in the past. The modular dual mobility acetabular cup, which can be fixed with screws, has a metal liner inserted therein, so there is a possibility that the concentration of metal ions in the blood may rise. Until now, studies on the concentration of metal ions in the blood after total hip arthroplasty using an modular dual mobility acetabular cup have been reported very rarely, and the results are also reported differently [4-7]. In addition, no prospective comparative study on blood metal ion concentrations after total hip arthroplasty using an modular dual mobility acetabular cup in elderly patients with femoral neck fractures has been reported. The release of metal ions due to metal corrosion or metal friction in the artificial joint is a rare phenomenon, but it can cause serious complications in the body. It has been suggested through case reports that it can cause abnormalities in the nervous system and cardiovascular system by increasing the concentration of metal ions in the body as well as bone complications such as osteolytic artificial joint relaxation pseudotumor around the artificial joint [5-7] , and a comparative analysis of the modular dual mobility acetabular cup with the conventional acetabular cup to see if there is any problem of metal ion rise in the body due to the release of metal ion concentration is a very important and meaningful study for both doctors and patients performing hip arthroplasty. In addition, it is expected that the medical and social contribution of this research will not be small, considering that the artificial prosthesis used as a material for metal-to-metal surface replacement surgery in the hip joint arthroplasty field was recalled a few years ago and caused a big wave around the world.

Matsen et al. defined significant elevation when Cobalt ≥ 1.6 mcg/L, based on previous literature that required revision for adverse local tissue reaction (ALTR). A guideline for follow-up of a metal artificial joint is attached as an appendix. Nam et al. (J Arthroplasty, 2016) reported that the frequency of patients with cobalt ion levels deviating from the normal reference values at 1 year after surgery was 4/26 (15.3%), MDM THA vs. 1/17 (5.9%) reported that it was Conventional THA. Matsen et al. did not specify the timing of the initial measurement of the ion concentration, but said that if abnormal values were observed, they were followed continuously every 6 months. Based on the previous literature that required revision for adverse local tissue reaction (ALTR), Cobalt ≥ 1.6 mcg/L was defined as significant elevation. As a result of following 100 patients, it was confirmed that the cobalt concentration was outside the normal range in 21 patients (21%), and a significant increase in the cobalt ion concentration of 1.6 mcg/L or more was reported in 9 patients (9%). And two of them had ALTR on MRI.

Metal ions can be released and the concentration of metal ions in the body can be increased in not only artificial joint replacement surgery using the assembled double movable acetabular cup but also in the solid acetabular cup. The acetabular cup and the femoral stem may be worn during joint movement due to the collision phenomenon, and if the acetabular cup screw is loosened or incorrectly inserted and corroded and worn, metal ions may be released along with the surrounding osteolysis.

The reason for performing randomization in this study is first, to ensure that the subject's characteristics do not affect the group to be assigned, so that the probability that each subject will receive surgery with which of the two substitutes is equally applied. , Second, in order to maximize the internal validity of the research results, to make the characteristics of the subjects to which the substitutes to be compared belong to be as similar as possible except for the substitutes assigned to them. Third, since statistical analysis was developed based on the theory of probability, The reason for randomizing the assignment of study subjects to the substitutions used is because it satisfies the prerequisites for applying statistical techniques to the analysis of research data.

Comparing and analyzing the difference in the concentration of metal ions in the blood through randomization is an important study that can confirm whether the difference in metal ion release can be caused by the difference in the binding mechanism between the two acetabular cups. It is an important complication after joint arthroplasty that can cause side effects and can cause harm to internal organs or revision surgery. Therefore, analyzing it is very important and meaningful research.

The purpose of this study was to compare the blood metal ion concentration in elderly patients after total hip arthroplasty using an modular dual mobility acetabular cup with the results of the conventional total hip arthroplasty patient group in a multicenter prospective study. In addition, we intend to compare clinical and radiological factors that are commonly evaluated during outpatient follow-up after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Over 60 years of age. Femoral neck fracture or hip joint disease. Garden stage III, IV
2. Comorbidities: American Society of Anesthesiology (ASA) grade III or less, Charlson comorbidity 6 points or less
3. Daily activity: UCLA score 4 or higher, Koval score 4 or lower
4. Including patients with neuromuscular disorder and cognitive impairment

Exclusion Criteria:

1. Revision arthroplasty
2. In case of factors other than fretting corrosion of the index arthroplasty that can cause an increase in serum metal ion level - In case of undergoing surgery using metal on other joints before this operation, vitamin B user
3. Patients with abnormal kidney function in which Blood urea nitrogen (BUN) and Cr are out of normal values
4. Pathologic fracture
5. If you have metabolic bone disorder, exclude osteoporosis (ex. Paraneoplastic syndrome, renal osteodystrophy, Vit D disorder, hormonal disorder)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Metal ion level | Baseline (pre op.), post op. 12 months
  Measurement of metal ion concentration in blood serum

SECONDARY OUTCOMES:
Change in Clinical measurement (Pain-visual analog scale) | Post op. 6 months, post op. 12 months, post op. 24 months
  Pain-visual analog scale
Change in Clinical measurement (Harris hip score) | Post op. 6 months, post op. 12 months, post op. 24 months
  Harris hip score
Change in Clinical measurement (Oxford hip score) | Post op. 6 months, post op. 12 months, post op. 24 months
  Oxford hip score
Change in Clinical measurement (UCLA score) | Post op. 6 months, post op. 12 months, post op. 24 months
  University of California at Los Angeles (UCLA) activity score
Change in Radiological measurement (Hip x-ray) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Acetabular cup inclination (degree)
Change in Radiological measurement (CT) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Anterior angle (degree, measured by computed tomography)
Change in Radiological measurement (Long leg x-ray) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Leg length difference (mm)
Post operative complication (Dislocation) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Dislocation or not
Post operative complication (Infection) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Infection or not
Post operative complication (Osteolysis) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Osteolysis or not
Post operative complication (Implant dissociation) | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Implant dissociation or not
Revision surgery | Baseline (immediate post op.), post op. 6 months, post op. 12 months, post op. 24 months
  Revision surgery or not

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin Kim, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- KoreaUGuroH, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No